CLINICAL TRIAL: NCT04668833
Title: Phase II Study of Autologous Lymphocyte Infusions After Radiation Therapy to Mitigate Radiation Induced Lymphopenia and Enhance Immune Reconstitution in Patients With Solid Tumor Malignancies
Brief Title: ALI Post Radiation Therapy in Patients With Lung and Esophageal Canter
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1164; NCI-2020-07836 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Autologous Lymphocyte Infusions) (Experimental): The purpose of this study is to determine the safety and preliminary efficacy of un-manipulated autologous lymphocyte infusion (ALI) using the patient's own lymphocytes collected using apheresis, and infused after the completion of radiation/chemoradiation.
  Interventions: Procedure: Autologous lymphocyte infusion (ALI)

INTERVENTIONS:
Procedure: Autologous lymphocyte infusion (ALI) — On the day after completing the last dose of radiation therapy, the patient will have an appointment scheduled in the Apheresis Unit for the infusion of unmunipulated cryopreserved cells. Patients will be pre medicated with acetaminophen (325-650 mg PO) and diphenhydramine (12.5-25 mg PO or IV) prior to infusion. Cells will be infused without a leukoreduction filter at a rate determined by cell volume.

SUMMARY:
The goal of this clinical research study is to learn if giving autologous lymphocyte infusions to patients who are receiving chemotherapy and radiation for non-small cell lung cancer or esophageal cancer is safe and effective.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and preliminary efficacy of un-manipulated autologous lymphocyte infusion (ALI) using the patient's own lymphocytes collected using apheresis, and infused after the completion of radiation/chemoradiation. Primary Objective To investigate the preliminary efficacy of autologous lymphocyte infusion (ALI) in improving the absolute lymphocyte counts in lung and esophageal cancer patients who had undergone chemo-radiation (CRT). Secondary Objectives

1. To evaluate the feasibility and safety of ALI in patients who had undergone chemoradiation.
2. To identify lymphocyte clonal populations in the tissue that are specific for tumor cells
3. To identify immune reconstitution in the peripheral blood shaped by ALI.
4. To conduct clonal analysis using T-cell receptor (TCR) sequencing from tumor and from peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically documented NSCLC or esophageal cancers Stage II-IVA disease where definitive chemoradiation is the standard of care Age 18

Exclusion Criteria:

Prior radiotherapy to the chest Life expectancy<6 months Any systemic therapy, aside from standard of care immunotherapy, that is planned to be administered prior to 6 weeks after ALI. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
To evaluate the absolute lymphocyte counts in lung and esophageal cancer patients who had undergone chemoradiation. (CRT) | Baseline to 6 weeks
  The primary outcome is the change between the two measures, i.e., absolute lymphocyte counts at week 6 (+/- 14 days) minus baseline ALC, referred as ALC change. Recently, we reviewed 755 patients with stage I-III esophageal carcinoma who received concurrent CRT with or without surgery in 2004-2015 [1]. The means of the absolute lymphocyte counts were 1,570 cells/µL (SD=610) and 980 cells/µL (SD=600) at based line and at the first follow-up visit post-CRT, respectively. We incorporate this clinical evidence in our sample size justification.

SECONDARY OUTCOMES:
To evaluate the feasibility of ALI in patients who had undergone chemoradiation. | Baseline to 6 weeks
  The number of patients who fail to complete the planned ALI treatment (i.e., inability to collect cell dose or receive cell infusion), will be counted and used as the summary of feasibility for this study. We will evaluate the feasibility of this study for future research and, it will be considered as feasible if less than 5 patients fail planned ALI treatment, while it will be stopped if 10 or more patients fail the planned ALI treatment during any time of the trial. The primary outcome of ALC will be summarized by means and standard deviations along with box-and-whisker plots.
To evaluate the safety of ALI in patients who had undergone chemoradiation. | Baseline to 6 weeks
  The method of Thall, Simon and Estey (1995) will be used for toxicity monitoring for this study. Denote the probability of toxicity by PT. We assume a priori, PT ~ beta (0.2, 1.8).
  We will stop the arm if Pr(PT> 0.1 | data)>0.80. That is, we will stop the arm for new patient enrollment if at any time during the study, we determine that there is more than 80% chance that the toxicity rate is more than 10%. This toxicity stopping rule will be applied starting from the 10th patient.

CONTACTS AND LOCATIONS:
Overall Officials: Gheath Al-Atrash, Principal Investigator — MD Anderson Cancer Center, Houston, Texas
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT04668833/ICF_000.pdf